CLINICAL TRIAL: NCT06441162
Title: A Pilot, Non-randomized, Single-site Clinical Study Investigating the Efficacy of Combined Therapy of Nebulized 3% Hypertonic Saline and Chest Percussion Therapy in Pediatric Patients With Acute Viral Bronchiolitis.
Brief Title: Efficacy Of Combined Nebulized Hypertonic Saline and Chest Percussion Therapy in Acute Viral Bronchiolitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-01357
Record Dates: First submitted 2024-05-29; First posted 2024-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Acute Bronchiolitis
Keywords: acute bronchiolitis; nebulized hypertonic saline; chest percussion therapy
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Nebulized Hypertonic Saline + Chest Percussion Therapy (Experimental): Participants with acute viral bronchiolitis will receive 3% nebulized hypertonic saline treatments combined with 3 minutes of chest percussion therapy. This will be administered every 6 hours.
  Interventions: Drug: Nebulized 3% sodium chloride solution; Device: Chest percussion cups
- Control Arm (No Intervention): Participants in the control arm will be analyzed via retrospective chart review; these participants will not be consented nor enrolled in the trial.

INTERVENTIONS:
Drug: Nebulized 3% sodium chloride solution — Standardized dose of nebulized 3% sodium chloride will be provided from 4 mL vial and administered be every 6 hours.
  Arms: Nebulized Hypertonic Saline + Chest Percussion Therapy
Device: Chest percussion cups — The chest percussion cup is a small, flexible cup made of vinyl that is used to provide gentle chest wall vibrations to assist with airway clearance and is utilized in patients of all ages with sputum production, such as those with acute bronchiolitis. Administered every 6 hours while on supplemental oxygen therapy.
  Other Names: MC-2247 Pediatric Manual Percussor Cup
  Arms: Nebulized Hypertonic Saline + Chest Percussion Therapy

SUMMARY:
This study will examine the efficacy of combined nebulized hypertonic saline with chest percussion therapy in patients age 0 to 24 months admitted to the general inpatient pediatrics unit with acute bronchiolitis. 3% nebulized hypertonic saline treatments combined with 3 minutes of chest percussion therapy will be administered every 6 hours of patients selected for the study.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study (experimental arm), an individual must meet all of the following criteria:

* Age 0 to 24 months
* Admitted to the general inpatient pediatrics unit
* Has a diagnosis of acute bronchiolitis
* Receiving supplemental oxygen support

Data collected for the control arm will be obtained via retrospective chart review for patients meeting the following inclusion criteria:

* Age 0 to 24 months
* Admitted to the general inpatient pediatrics unit
* Has a diagnosis of acute bronchiolitis
* Receiving supplemental oxygen support

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Admitted to the pediatric intensive care unit
* Has an underlying pre-existing condition that may affect the respiratory system (includes bronchopulmonary dysplasia, reactive airways disease, asthma, restrictive lung diseases, other chronic lung diseases, etc.)
* Has other comorbid conditions upon admission that may affect the respiratory system (includes pneumonia or other bacterial or fungal lung infections, acute exacerbation of reactive airways disease, acute exacerbation of asthma, pulmonary edema, pleural effusion, etc.)
* Has an absolute contraindication to nebulized 3% hypertonic saline, for example, a history of an allergic or anaphylactic reaction
* Is receiving other respiratory treatments such as bronchodilator treatments (i.e. albuterol or levalbuterol)
* Is receiving other adjuvant therapy such as antibiotics, antivirals, glucocorticoids, corticosteroids, or diuretics

A potential study subject in the control arm via retrospective chart review who meets any of the following criteria will be excluded from this study:

* Admitted to the pediatric intensive care unit
* Has an underlying pre-existing condition that may affect the respiratory system (includes bronchopulmonary dysplasia, reactive airways disease, asthma, restrictive lung diseases, other chronic lung diseases, etc.)
* Has other comorbid conditions upon admission that may affect the respiratory system (includes pneumonia or other bacterial or fungal lung infections, acute exacerbation of reactive airways disease, acute exacerbation of asthma, pulmonary edema, pleural effusion, etc.)
* Has an absolute contraindication to nebulized 3% hypertonic saline, for example, a history of an allergic or anaphylactic reaction
* Is receiving other respiratory treatments such as bronchodilator treatments (i.e. albuterol or levalbuterol)
* Is receiving other adjuvant therapy such as antibiotics, antivirals, glucocorticoids, corticosteroids, or diuretics

Ages: 0 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Actual)
Dates: Start 2024-07-15 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
Length of Hospital Stay | Up to time of discharge (Approximately 1-5 days on average)
  Measured in days from from time of admission to the general inpatient pediatrics unit until time of discharge from the general inpatient pediatrics unit.
Time on Supplemental Oxygen Support | Up to time of discharge (Approximately 1-5 days on average)
  Measured in days from from time of admission to the general inpatient pediatrics unit until time of discharge from the general inpatient pediatrics unit.

SECONDARY OUTCOMES:
Average Respiratory Rate | Up to time of discharge (Approximately 1-5 days on average)
  Assessed every 4 hours and as needed in addition.
Average Heart Rate | Up to time of discharge (Approximately 1-5 days on average)
  Assessed every 4 hours and as needed in addition.
Average Pulse Oximetry Reading | Up to time of discharge (Approximately 1-5 days on average)
  Assessed every 4 hours and as needed in addition.
Number of Caregivers who Rate Child's Response as "Improved" | Time of discharge (Approximately 1-5 days on average)
  Caregivers will be given a survey in which they will rate their child's overall response following the treatments as "Improved," "Unchanged," or "Worsened."
Number of Physicians who Rate Child's Response as "Improved" | Time of discharge (Approximately 1-5 days on average)
  Caregivers will be given a survey in which they will rate their child's overall response following the treatments as "Improved," "Unchanged," or "Worsened."

CONTACTS AND LOCATIONS:
Overall Officials: Tuan Nguyen, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, Mineola, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: Tuan Nguyen tuan.nguyen@nyulangone.org 405-535-7093 The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to tuan.nguyen@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.